CLINICAL TRIAL: NCT03633188
Title: Stool Biobanking and Impact of Antimicrobials on the Gut Microbiota in Patients With Bone and Joint Infection
Acronym: GUMIBONE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study had to be stopped because the period of the Financial contract was over
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: University of Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0652; 2017-A02813-50 (Other: ANSM)
Record Dates: First submitted 2018-07-17; First posted 2018-08-16 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Infection, Bacterial
Keywords: Bone and Joint Infections (BJI); gut dysbiosis; antimicrobial resistance; antibiotic resistance gene; mobile genetic elements
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated by antibiotherapy (Experimental): 35 Patients treated by antibiotherapy for acute and subacute post-operative implant-associated BJI infections and among them 10 patients with Staphylococcus. aureus treated with antibiotics as part of their standard treatment procedure for metagenomic procedure.
  Interventions: Biological: Patients treated by antibiotherapy

INTERVENTIONS:
Biological: Patients treated by antibiotherapy — Biological samples (stool, blood, swabs) will be collected :
  * Blood sampling (12 ml) at baseline (week 0) at the end of treatment (W6/W24),and 15 days after antibiotherapy stop (optional) (W8/W26),
  * Feces collection at baseline (week 0) during antibiotic treatment (W2), at the end of treatment (W6/W24),15 days after antibiotherapy stop (W8/W26), and W26 after baseline
  * Swab samples (nasal and rectal) at baseline at week 0 and at the end of treatment (W6/W24),

SUMMARY:
Bone and joint infections (BJI) is a public health issue in industrialized countries.

Implant-associated BJI, are complex hospital-acquired infections and eradication of the pathogen is challenging in such patients.

A prolonged antimicrobial therapy is usually required from 6 weeks to 3 months, but some patients are eligible to several years of treatment and most of patients report gastrointestinal troubles, such as nausea and mild to severe diarrhea (but very few developed C. difficile diarrhea).

Moreover, the host gut microbiota is probably largely affected in abundance, richness and diversity. Indeed, it is known, that few days of antibiotics are sufficient to induce significant alterations of the gut microbiota, also called dysbiosis.

Severe dysbiosis, which is potentially irreversible and associated with a definitive shift in the gut microbiota metabolism and host homeostasis, may lead to and/or promote a large panel of severe diseases such as Clostridium difficile infection, diabetes mellitus, obesity, inflammatory bowel disease (IBD), cirrhosis, neurological disorders and cancer. It may also be associated with BJI recurrence and then impact global health costs.

The main objective of this study is to constitute biobanking of stools and perform DNA sequencing of the gut microbiota in patients with acute or sub-acute implant-related Bone and Joint Infection (BJI), caused by Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing, able to understand and comply to the protocol requirement
2. More than 18-years-old
3. Subject with suspicion of implant-related BJI within 3 months after surgery and treated by antibiotherapy for a maximal duration of six months
4. Subject signed Inform Consent Form
5. Contraception for women of childbearing age

Exclusion Criteria:

1. Pregnancy
2. Severe disease with a life expectancy < 3months
3. Any antibiotherapy treated all diseases in the 14 days before inclusion
4. Guardianship, curatorship patients
5. Patient non-affiliated to health care system
6. Patient under the power of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
change in the gut microbiota after treatment | from baseline to week 26
  stools will be collected to perform DNA sequencing of the gut microbiota in patients with acute or sub-acute implant-related Bone and Joint Infection (BJI), caused by Staphylococcus aureus.
  Stools will be collected at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.

SECONDARY OUTCOMES:
Assessment of the evolution of intensity of Diarrheic Symptoms | from baseline to week 8 or week 26
  intensity of diarrheic symptoms will be collected at baseline, at the end of treatment (Week 6 or Week 24) and 15 days after antibiotic stop (Week 8 or Week 26)
Assessment of the evolution of frequency of Diarrheic Symptoms | from baseline to week 8 or week 26
  frequency of diarrheic symptoms will be collected at baseline, at the end of treatment (Week 6 or Week 24) and 15 days after antibiotic stop (Week 8 or Week 26)
Quantity of rectal acquisition of Multi Drug Resistance (MDR) bacteria under antibiotics measured by classic culture and quantification culture methods | at week 6 or week 24
  classic culture and quantification culture methods determined by microbiology analysis of the feces.
  Feces will be collected at baseline and at the end of treatment
gut dysbiosis measured by Next Generation Sequencing (NGS) | from baseline to week 26
  Stools will be collected at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.
  Microbiota sequencing will be done after DNA extraction. Composition of the microbiota will be screened in feces samples using the shotgun sequencing method to establish a total picture of the gut composition and diversity as well as evolution of the microbiome.
severe post-antibiotic dysbiosis (SPAD) measured by Next Generation Sequencing (NGS) | from baseline to week 26
  Severe Post-Antibiotic Dysbiosis lead to irreversible change in gut microbiota status and systemic consequences for the host.
  Stools will be collected at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.
Identification of markers of the gut dysbiosis (inflammatory proteins) measured by Elisa techniques | from baseline to week 26
  ELISA techniques will be used to determine the concentration of 3 specific inflammatory stool epithelium proteins: zonulin, calprotectin and neopterin.
  Stools will be collected at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.
Analysis of impact of Bone and Joint Infection on health-related quality of life in patients by EQ5D5L questionnaires | from baseline to week 26
  EQ-5D questionnaire has 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression". All dimensions are described by 5 (EQ-5D-5L) problem levels corresponding to patient response choices.
  Questionnaire will be completed at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.
Analysis of impact of Bone and Joint Infection on health-related quality of life in patients by EQ5D3L questionnaire | from baseline to week 26
  EQ-5D questionnaire has 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression". All dimensions are described by 3 (EQ-5D-3L) problem levels corresponding to patient response choices. In France, only the EQ-5D-3L has been validated, not yet the EQ-5D-5L which has only been translated.
  Questionnaire will be completed at baseline, during antibiotic treatment (Week 2), at the end of treatment (Week 6 or Week 24),15 days after antibiotherapy stop (Week 8 or Week 26), and W26 after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Hôpital de la Croix Rousse-Service de chirurgie orthopédique, Lyon
  - Hôpital de la Croix Rousse-Service des Maladies Infectieuses et Tropicales, Lyon
  - Centre Hospitalier Lyon Sud-Service de Chirurgie Orthopédique, Pierre-Bénite
  - Centre Hospitalier Lyon Sud-Service des maladies infectieuses, Pierre-Bénite